CLINICAL TRIAL: NCT04125238
Title: Reinforcer Pathology 1A: Increasing the Temporal Window
Brief Title: Increasing the Temporal Window in Individuals With Alcohol Use Disorder
Acronym: RP1A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); McMaster University (Other); Arizona State University (Other); Carilion Clinic (Other); University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RP1A / 20-015 / 22-358; R01AA027381-01A1 (NIH)
Record Dates: First submitted 2019-10-09; First posted 2019-10-14 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use Disorder
Keywords: Delay Discounting; Behavioral Economic Demand; Episodic Future Thinking; Self-Administration; Functional MRI; Alcohol Craving
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episodic Future Thinking (EFT) (Experimental): Participants will generate positive future events they are looking forward to at five time points in the future (1 day, 1 week, 1 month, 3 months, 1 year, 5 years, and 25 years). Participants will be reminded of these events using cues throughout the study and instructed to think about these cues as they make their decisions.
  Interventions: Behavioral: Episodic Future Thinking
- Control Episodic Thinking (CET) (Sham Comparator): Participants will generate positive recent past events that have happened to them at five time points in the recent past (last night from 7pm-10pm, yesterday between 4pm-7pm, yesterday between 1pm-4pm, yesterday from 10am-12pm, yesterday between 7am-10am, the night before last between 7pm-10pm, and evening before last between 4pm-7pm). Participants will be reminded of these events using cues throughout the study and instructed to think about these cues as they make their decisions.
  Interventions: Behavioral: Control Episodic Thinking

INTERVENTIONS:
Behavioral: Episodic Future Thinking — Participants will generate descriptions of vivid positive future events.
  Other Names: EFT
  Arms: Episodic Future Thinking (EFT)
Behavioral: Control Episodic Thinking — Participants will generate descriptions of vivid positive recent past events.
  Other Names: CET
  Arms: Control Episodic Thinking (CET)

SUMMARY:
Episodic future thinking (EFT) is based on the new science of prospection, which was first identified in a Science publication in 2007 and refers to pre-experiencing the future by simulation. Considerable evidence suggests that prospection is important for understanding human cognition, affect, motivation, and action. Individuals with damaged frontal areas, as well as individuals with alcohol use disorder (AUD), show deficits in planning prospectively. One systematic method to engender prospection is via EFT. EFT, as applied in our prior studies and in this proposal consists of having participants develop positive plausible future events that correspond to several future time frames (e.g., 2 weeks, 1 month, 3 months etc). For each of these timeframes participants are asked to concretize the events (e.g., What are you doing? Who will be there? What will you see, hear, smell, and feel?). We and others have used EFT to decrease delay discounting (DD) in individuals with AUD and smokers, as well as normal weight, overweight, and obese populations when compared to the control condition, control episodic thinking (CET). Consistent with reinforcer pathology, EFT also reduces alcohol valuation in the purchase task among individuals with AUD. However, no study to date has examined whether EFT reduces alcohol self-administration in the laboratory. Moreover, the neural correlates of EFT in AUD are also unknown. In these studies, we propose to test an intervention, EFT, which we hypothesize will decrease reinforcer pathology measures in a bar-like setting in the laboratory; that is, EFT will decrease delay discounting, as well as alcohol self-administration, demand, and craving compared to a control episodic thinking (CET) condition. Moreover, we hypothesize EFT will enhance activation in brain regions associated with prospection (e.g., hippocampus and amygdala) and the executive decision system (e.g., DLPFC). We will also examine the effect of EFT on real-world drinking.

DETAILED DESCRIPTION:
In study 1, participants will be randomly assigned to experimental or control groups, stratified by AUDIT scores, SES, age and sex. Based on our 8 years of experience recruiting this population, we expect approximately 66% retention among eligible participants. Therefore, we will enroll approximately 107 participants in order to conclude with 64 completers. Participants will complete: a baseline assessment (S1), an alcohol self-administration session (S2 or S3), an fMRI session (S2 or S3). The alcohol self-administration session and the fMRI session will be completed in counterbalanced order. At the beginning of S2 and S3, participants in both groups will be prompted to generate positive events and related cues through a researcher-administered interview-based questionnaire. EFT group participants will be asked to think about and describe the most positive event that could realistically happen at each of 7 delays in the future (1 day, 1 week, 1 month, 3 months, 1 year, 5 years, and 25 years). In contrast, participants randomized to the CET condition, will be asked to think about and describe the most positive event that occurred at each of 7 time points from the recent past (last night from 7pm-10pm, yesterday between 4pm-7pm, yesterday between 1pm-4pm, yesterday from 10am-12pm, yesterday between 7am-10am, the night before last between 7pm-10pm, and evening before last between 4pm-7pm). For each time point, the participant will be asked to integrate the event and sensory information into concise textual and/or auditory cues to be used in subsequent behavioral tasks. Cue generation will occur prior to both self administration and fMRI sessions (S2 and S3) to maximize the relevancy of cues at both sessions.

In study 2, participants will complete two sessions and undergo a one-week baseline monitoring phase where they provide breath samples to assess for recent alcohol use and report their drinks per day. Following this baseline period, participants will complete an fMRI then be randomized to either the EFT or Control group. Participants will then complete two weeks of monitoring, where they provide a breath sample three times a day and report the number of drinks they consumed. Participants will then come back to the lab to generate new EFT/CET cues, then complete two more weeks of monitoring. After conclusion of the second intervention period, participants will complete a post intervention session and then a one month follow up one month after study completion.

ELIGIBILITY:
Inclusion Criteria:

* High-risk or harmful drinking (measured by AUDIT)
* 21-65 years of age
* Desire to quit or cut down on their drinking, but do not have proximate plans to enroll in treatment for AUD during the study period
* Report as one of their top three preferred drinks a beverage appropriate for the alcohol self-administration task (Study 1)

Exclusion Criteria:

* Moderate to severe DSM-5 criteria for substance-use disorders other than alcohol, nicotine, and/or marijuana
* Current diagnosis of any psychotic disorder
* History of seizure disorders or traumatic brain injury
* Contraindication for participation in the self-administration (Study 1) or MRI sessions (Studies 1 and 2)
* Current pregnancy or lactation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M LaConte, PhD, Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will adhere to all NIH requirements regarding data sharing. Participant data collected in this project will be de-identified and made available on a shared secured data repository. We will also share the analysis results. As part of this process, all investigators will be required to agree to the following conditions: 1) will adhere to the reporting responsibilities; 2) will not redistribute the data beyond the requesting individual and named collaborators; 3) will give appropriate acknowledgement; 4) will not use the data for commercial purposes; and 5) will obtain appropriate ethical approvals.
  Results from research conducted will be shared and disseminated, including: regular project meetings, annual meetings, symposia, workshops, and/or conferences for related groups. Manuscripts will be written and submitted for publication in peer-reviewed journals/conferences, following the NIH Public Access Policy guidelines. All necessary ethical approvals will be obtained.
Time Frame: Data will be made available upon request after dissemination of results.
Access Criteria: Data requests will be reviewed by the principal investigator and data will be shared with the expectation of acknowledgment of funding source and primary study team.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study 1: 38 participants signed consent and enrolled in Study 1. Study 2: 116 participants signed consent and enrolled in Study 2. Two of those participants were pilots. Furthermore, randomization occurred after a 7-day baseline period, and only participants who met the study's baseline criteria were invited to continue and assigned to groups. Therefore, out of the 114 non-pilot participants enrolled, 64 were randomized. Only randomized participants (n=64) are included in the numbers below.
Groups:
- Episodic Future Thinking (EFT) - Study 1; Episodic Future Thinking (EFT) - Study 2: Participants will generate positive future events they are looking forward to at five time points in the future (1 day, 1 week, 1 month, 3 months, 1 year, 5 years, and 25 years). Participants will be reminded of these events using cues throughout the study and instructed to think about these cues as they make their decisions.
  Episodic Future Thinking: Participants will generate descriptions of vivid positive future events.
- Control Episodic Thinking (CET) - Study 1; Control Episodic Thinking (CET) - Study 2: Participants will generate positive recent past events that have happened to them at five time points in the recent past (last night from 7pm-10pm, yesterday between 4pm-7pm, yesterday between 1pm-4pm, yesterday from 10am-12pm, yesterday between 7am-10am, the night before last between 7pm-10pm, and evening before last between 4pm-7pm). Participants will be reminded of these events using cues throughout the study and instructed to think about these cues as they make their decisions.
  Control Episodic Thinking: Participants will generate descriptions of vivid positive recent past events.
Period: Overall Study
Arm/Group | Episodic Future Thinking (EFT) - Study 1 | Control Episodic Thinking (CET) - Study 1 | Episodic Future Thinking (EFT) - Study 2 | Control Episodic Thinking (CET) - Study 2
Started (For Study 2, 116 participants signed a consent form, but 2 were pilot participants, and out of the 114 remaining, only 64 met the baseline criteria and were randomized for one of the conditions.) | 20 | 18 | 34 | 30
Completed | 16 | 12 | 28 | 24
Not Completed | 4 | 6 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Episodic Future Thinking (EFT) - Study 1 | Control Episodic Thinking (CET) - Study 1 | Episodic Future Thinking (EFT) - Study 2 | Control Episodic Thinking (CET) - Study 2 | Total
Number analyzed (Participants) | 20 | 18 | 34 | 30 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (8.95) | 42.4 (12.96) | 39.74 (13.52) | 35.7 (12.35) | 39.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 12 | 13 | 39
  Male | 14 | 10 | 22 | 17 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 2 | 5
  Not Hispanic or Latino | 19 | 18 | 32 | 28 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Delay Discounting (DD) Rates (Studies 1 and 2)
Description: DD rates were measured using an adjusting amount task where participants were presented with hypothetical choices between smaller immediate or larger later amounts of money after a range of delays (1 day-25 years). Individual indifference points were calculated for each delay and then used to estimate DD rates for each participant using Mazur's (1987) equation: V = A/(1+kD), where V is the value of the indifference point, A is the amount of the larger delayed reward, k is the discounting rate, and D is the delay. Discounting rates (k) were then natural-logarithmically transformed (ln(k)). Higher ln(k) indicates steeper discounting and greater reward devaluation with increases in delay, while a lower ln(k) reflects shallower discounting and less reward devaluation with increases in delay.
  Change in ln(k) will be compared within-subjects between S1 and S2, AND between S1 and S3.
Time Frame: Pre-intervention (S1; baseline measures; Day 1), Post 1st cue generation: S2 (occurs up to 7 days post S1 in Study 1 and 2-3 weeks post S1 in Study 2), and Post 2nd cue generation: S3 (occurs up to 7 days post S2 in Study 1 and 2 weeks post S2 in Study 2)
Population: Only participants who completed both cue generation sessions were included in the analyses.
Measure: Mean (Standard Error); unit: ln(K-value)
Arm/Group | Episodic Future Thinking (EFT) - Study 1 | Control Episodic Thinking (CET) - Study 1 | Episodic Future Thinking (EFT) - Study 2 | Control Episodic Thinking (CET) - Study 2
Number analyzed (Participants) | 16 | 11 | 31 | 26
ln(K-value)
  Pre-intervention | -5.33 (0.44) | -6.03 (0.41) | -4.94 (0.44) | -5.79 (0.49)
  Post 1st cue gen | -6.72 (0.65) | -5.94 (0.55) | -6.41 (0.39) | -5.1 (0.45)
  Post 2nd cue gen | -6.61 (0.50) | -5.75 (0.38) | -6.54 (0.40) | -5.28 (0.59)

2. Primary Outcome: Intensity of Alcohol Demand (Study 2)
Description: Participants completed a hypothetical Alcohol Purchase Task in which they indicated how many drinks they would purchase at different prices ($0 to $80 per drink). The number of drinks purchased at $0 was used to calculate the intensity of demand. Changes in intensity of alcohol demand were compared within-subjects between S1 and S2, AND between S1 and S3.
Time Frame: Pre-intervention (S1; baseline measure; Day 1), Post 1st cue generation, (S2; approximately 2 weeks post S1), and Post 2nd cue generation (S3; approximately 2 weeks post S2 and 4 weeks post S1)
Population: Only participants who completed both cue generation sessions were included in the analyses.
Measure: Mean (Standard Deviation); unit: Drinks
Arm/Group | Episodic Future Thinking (EFT) - Study 2 | Control Episodic Thinking (CET) - Study 2
Number analyzed (Participants) | 31 | 26
Drinks
  S1 | 11.19 (5.98) | 15.04 (9.79)
  S2 | 11.22 (7.23) | 14.27 (6.81)
  S3 | 10.87 (7.17) | 14.65 (10.14)

3. Primary Outcome: In-Laboratory Alcohol Consumption (Study 1)
Description: The number of alcoholic beverages purchased/consumed during the self-administration session will be recorded. The average number of drinks consumed will be compared between groups.
Time Frame: Self-Administration session will occur at either Session 2 or Session 3 based on counterbalance assignment. S2 occurs up to 7 days post S1 and S3 occurs up to 7 days post S2.
Population: Only participants who completed the Self-Administration session were included in the analysis.
Measure: Mean (Standard Deviation); unit: Drinks
Arm/Group | Episodic Future Thinking (EFT) | Control Episodic Thinking (CET)
Number analyzed (Participants) | 16 | 12
Drinks | 4.81 (2.81) | 5.25 (3.22)

4. Primary Outcome: fMRI Hyper-connectivity Decrease During Delay Discounting (Study 1)
Description: Measured using fMRI during delay discounting task. Whole-brain PPI analysis of right DLPFC between EFT and CET participants. We examined the number of participants whose Right DLPFC was negatively correlated with their Left DLPFC after the intervention. We hypothesize that AUD leads to hyperconnectivity (positive correlations) between these two regions as a compensatory decision-making mechanism, and that EFT should reduce or reverse this connectivity relationship
Time Frame: fMRI session occurred at either Session 2 or Session 3 based on counterbalance assignment. S2 occurred up to 7 days post S1 and S3 occurred up to 7 days post S2.
Population: Only participants who completed the fMRI scan and showed acceptable motion and no artifacts were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Episodic Future Thinking (EFT) | Control Episodic Thinking (CET)
Number analyzed (Participants) | 15 | 9
Participants | 14 | 0

5. Primary Outcome: fMRI Hyper-connectivity Decrease During Alcohol Purchase Task (Study 1)
Description: Measured using fMRI during the alcohol purchase task. Whole-brain PPI analysis of right DLPFC between EFT and CET participants. We examined the number of participants whose Right DLPFC was negatively correlated with their Left DLPFC after the intervention. We hypothesize that AUD leads to hyperconnectivity (positive correlations) between these two regions as a compensatory decision-making mechanism, and that EFT should reduce or reverse this connectivity relationship
Time Frame: as for outcome 4
Population: Only participants who completed the fMRI scan and showed acceptable motion and no artifacts were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Episodic Future Thinking (EFT) | Control Episodic Thinking (CET)
Number analyzed (Participants) | 15 | 9
Participants | 0 | 0

6. Primary Outcome: Change in Alcoholic Drinks Per Day (Study 2)
Description: Participants self-reported the number of drinks consumed per day via a mobile app during the first five weeks of the study. The first week measured baseline drinking (Pre-intervention), weeks 2-3 measured drinking after the first cue generation (Post 1st cue generation), and weeks 4-5 measured drinking after the second cue generation (Post 2nd cue generation) The number of drinks per day was compared within-subjects and between groups (EFT and CET).
Time Frame: Daily during Pre-intervention (week 1); Post 1st cue generation (weeks 2-3); and Post 2nd cue generation (weeks 4-5).
Population: Only participants who completed the entire intervention (all 5 weeks) were included in this analysis.
Measure: Mean (Standard Error); unit: Drinks/day
Arm/Group | Episodic Future Thinking (EFT) | Control Episodic Thinking (CET)
Number analyzed (Participants) | 30 | 24
Drinks/day
  Pre-Intervention | 5.6 (0.41) | 5.3 (0.42)
  Post 1st cue generation | 5.0 (0.42) | 4.9 (0.43)
  Post 2nd cue generation | 4.3 (0.37) | 5.4 (0.62)

ADVERSE EVENTS:
Time Frame: During study participation (up to 14 days in Study 1, and 35 days in Study 2)
Description: Withdrawal symptoms were measured via self-report at the beginning of each session.
Arm/Group | Episodic Future Thinking (EFT) - Study 1 | Control Episodic Thinking (CET) - Study 1 | Episodic Future Thinking (EFT) - Study 2 | Control Episodic Thinking (CET) - Study 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18 | 0/34 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/34 | 0/30
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/34 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04125238/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04125238/SAP_001.pdf